CLINICAL TRIAL: NCT02860312
Title: Effects of One Year Perdialytic Physical Activity on Aerobic Capacities and Quality of Life in Hemodialysis Patients
Brief Title: Long Term Physical Activity for Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AURA Sante (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AURAS; ID-RCB 2015-A0031-48 (Other: CPP Clermont Ferrand)
Record Dates: First submitted 2016-07-14; First posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: End Stage Renal Disease on Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercisers (Active Comparator): Intradialytic exercise on stationary bicycles
  Interventions: Behavioral: Intradialytic exercise on stationary bicycles
- Non Exercisers (Placebo Comparator): No intradialytic exercise
  Interventions: Behavioral: Non-exercising group

INTERVENTIONS:
Behavioral: Intradialytic exercise on stationary bicycles — Patients are exercising for 30-60 min during dialysis on an Rated Perceived Exertion (RPE) Scale between 12 and 14
  Arms: Exercisers
Behavioral: Non-exercising group — Patients are having their usual physical activity
  Arms: Non Exercisers

SUMMARY:
Patients on chronic hemodialysis present severe physical dysfunctioning associated with a significant reduction of their muscle mass. These two parameters are associated with increased morbidity and mortality along with deconditioning and poor quality of life. There are several studies- usually short term, single center uncontrolled and underpowered- that have shown a significant improvement of the physical, metabolic and dialytic parameters.

There are only few studies that have measured the impact of a long term intradialytic exercise intervention on a supervised manner. This is a multi-center controlled study examining the effects of intradialytic cycling on parameters of physical functioning, body composition, cardiovascular and nutritional status, immunological status and quality of life in a group of clinically stable hemodialysis patients

DETAILED DESCRIPTION:
General Context Chronic Kidney Patients (CKD) live a sedentary life. Sedentarity and Sarcopenia worsen during the evolution of CKD with numerous cardiovascular diseases, infectious and other comorbidities. Inactivity may activate and amplify the inflammatory process, hypercoagulability, malnutrition, invoking a vicious circle of further inactivity and deconditioning.

These populations have a very low physical activity profile due to important tiredness, perturbed general condition and bad adaptation in effort. The patients with cardiovascular problems have additional limitations due to breathlessness associated with congestive cardiac failure and intermittent claudication due to peripheral arteriopathy. At the dialysis stages the tiredness is accentuated after the hemodialysis sessions. The days off dialysis are rarely used for practicing a physical activity.

The deconditioning along with the reduction of the physical activity are leading to a de-socializing progressing in the course of the chronic renal failure. In that way the patient feels more and more isolated with a serious eventual impact on the nutrition status and his quality of life.

Regular physical activity in this population of patients is exerting beneficial effects on insulin resistance, inflammation, dialysis efficiency, nutrition and arterial pressure. It may also reduce the intradialytic hypotensive episodes and improve quality of life, without side effects.

The objective of this study is to investigate an improvement of the physical functioning associated with a reprogramming of the autonomous nervous system, a reduction of the pro-inflammatory factors with a reduction of the insulin resistance (reduction of the metabolic syndrome), along with improvements on the immune system functioning for hemodialysis patients participating on a one year intradialytic physical activity program.

Principal objective :

The principal aim of the present study is to show the efficacy of intradialytic physical activity on functional capacity with the sit-to-stand test in 60 seconds (STS60) and the time to perform 5 complete sit-to-stand movements (STS5) along with a 6 minutes' walk test (6MWT).

Secondary objectives :

The secondary objectives are the amelioration of parameters associated with cardiovascular, sympathetic or autonomous nervous system, immune, nutritional, metabolic and inflammatory outcomes among with quality of life.

This is a multicenter, controlled randomized trial

Study description:

Inclusion of patients willing to participate in the study, and consequently their randomization in 2 groups.

The intervention group will benefit from a supervised physical activity during the dialysis session and the other group will carry on with his usual physical activities and have the same tests before and after the trial without undergoing a supervised intradialytic physical activity program

Primary judgment criteria :

The principal criteria will be the effect of an aerobic training program with a warming up phase, followed by 30 minutes of intradialytic cycling on 55% of the VO2max, 3 times a week.

The primary judgement criteria will be the improvement of the Sit-to-stand test in 60 seconds (STS60) and the time to complete 5 sit-to stand movements (STS5) as well as the 6 minutes' walk test (6MWT) from T0 (before the training program) to T12 (12 months after the start of the training period)

Secondary criteria:

* Quality of life parameters evaluated from the questionaries SF36 (The Short Form (36) Health Survey), Borg scale, EVA.
* Physical activity levels: IPAQ (international physical activity questionary).
* Body composition (Fat mass, lean mass, bone mineral density, estimation of the muscular mass) with DEXA (dual-energy x-ray absorptiometry).
* Cardiovascular parameters : Cardiac echography, doppler of the carotid arteries and the lower extremity arteries, 24h cardiac rhythm exploration
* Immune parameters: leucocyte subpopulation functioning
* Nutritional and metabolic parameters: weight, BMI, albumin, pre-albumin, pre- and post-dialytic serum urea and creatinine levels, nPCR (normalised Protein catabolic Rate).
* Inflammatory parameters :(Interleucin) IL1 bêta, IL6, IL8, IL-10, TNF alpha (Tumor necrosis factor alpha), CRP (C reactive protein)
* Dialysis parameters : Kt/v, anemia control : Hemoglobin (Hb), MCV (mean corpuscular volume), ferritin, erythropoetin dosage (EPO).
* Number, etiology and duration of hospitalisations
* Survival in 1 year

Number of participants : 100, ie 50 per group

Layout of the study :

Inclusion of the patient, evaluations at the start of the study protocol, at 6 months and at the end -12 months (M0, M6, M12).

Benefits and risks of this study :

Improvement of functional aerobic capacity, inflammatory status and quality of life. Improvements on the state of pain, autonomy, augmentation of the lean mass with conservation of the muscular mass for the lower extremities and reduction of the total fat mass are expected as well as improvement of the nutritional status, dialysis parameters, anemia control.

The risks are of cardiovascular origin: a possible decompensation of coronary artery disease, peripheral artery disease, taking into consideration that all patients benefit from echo doppler arterial control before the start of the study.

Regular Perdialytic Activity during Dialysis is practiced in AURA Auvergne (Association pour l'Utilisation du Rein Artificiel Santé) since 2 years; there has been no secondary vascular problem associated with the supervised physical activity. Nevertheless, rare tendon problems or articular and muscular pains could be possible on the course of the study

ELIGIBILITY:
Inclusion Criteria:

* Consenting active hemodialysis patients since at least 6 months aged between 20 and 90 y.o.

Exclusion Criteria:

* Unstable angina,
* severe left ventricular dysfunction,
* Ejection fraction < 30%,
* severe peripheral arterial disease,
* lower extremity amputation,
* impossibility of physical effort: pain, uncontrolled bone/muscular disease,
* participation on another study.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Improvement of the distance covered after walking for 6 minutes (6 minutes walk test) | 12 months
  The principal aim of the present study is to show the efficacy of intradialytic physical activity on the improvement of the physical capacity of the patients assessed with the 6 minutes walk test ((6MWT)

SECONDARY OUTCOMES:
Quality of life parameters 1 | 12 months
  Quality of life parameters evaluated from the questionnaire SF36 QD
Quality of life parameters 2 | 12 months
  Quality of life parameters evaluated from the questionnaire Borg scale
Quality of life parameters 3 | 12 months
  Quality of life parameters evaluated from the EVA scale
Physical activity levels | 12 months
  Physical activity levels from the questionnary IPAQ (international physical activity questionnairy)
Body composition | 12 months
  Body composition (Fat mass, lean mass, bone mineral density, estimation of the muscular mass) with DEXA ccanning and bioimpendance
Cardiovascular parameters | 12 months
  Cardiovascular parameters : Cardiac echography, echodoppler of the carotid arteries and the lower extremity arteries, 24h cardiac rythm exploration
Immune parametres | 12 months
  Immune parametres: leucocyte subpopulation fonctioning
Nutritional and metabolic parameters 1 | 12 months
  BMI
Nutritional and metabolic parameters 2 | 12 months
  serum albumin levels
Nutritional and metabolic parameters 3 | 12 months
  serum prealbumin levels
Nutritional and metabolic parameters 4 | 12 months
  pre and post dialytic serum urea levels
Nutritional and metabolic parameters 5 | 12 months
  pre and post dialytic serum creatinine levels
Nutritional and metabolic parameters 6 | 12 months
  nPCR (normalised Protein Catabolic Rate)
inflammatory parameters 1 | 12 months
  IL1 bêta
inflammatory parameters 2 | 12 months
  IL6
inflammatory parameters 3 | 12 months
  IL8
inflammatory parameters 4 | 12 months
  IL-10
inflammatory parameters 5 | 12 months
  TNF alpha
inflammatory parameters 6 | 12 months
  CRP
Dialysis parameters | 12 months
  Kt/V
Anemia control 1 | 12 months
  Hemoglobin (Hb)
Anemia control 2 | 12 months
  MCV (mean corpuscular volume)
Anemia control 3 | 12 months
  Ferritine
Anemia control 4 | 12 months
  Erythropoetine dosage (EPO).
Number of hospitalisations | 12 months
  Number of hospitalisations
Duration of hospitalisations | 12 months
  Duration of hospitalisations
Survival | 12 months
  Survival in one year
Improvement of Sit to Stand test in 60 seconds (STS60) | 12 months
  The physical capacity of the patients assessed with the number of cycles performed during a sit-to-stand test in 60 seconds (STS60).
Improvement of the time needed to perform 5 Sit to Stand cycles (STS5) | 12 months
  Time needed to perform 5 Sit to Stand cycles (STS5)

IPD SHARING:
Plan to Share IPD: No